CLINICAL TRIAL: NCT00542984
Title: Comparison of Teriparatide and Calcitonin in the Treatment of Postmenopausal Women With Osteoporosis
Brief Title: Comparison Medications in the Treatment of Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6680; B3D-KL-GHCC
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide; salmon calcitonin; Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): teriparatide 20 micrograms/day subcutaneous
  Interventions: Drug: teriparatide 20 micrograms/day subcutaneous
- B (Active Comparator): salmon calcitonin 100 IU/day subcutaneous
  Interventions: Drug: salmon calcitonin 100 IU/day subcutaneous

INTERVENTIONS:
Drug: teriparatide 20 micrograms/day subcutaneous
  Other Names: LY333334
  Arms: A
Drug: salmon calcitonin 100 IU/day subcutaneous
  Arms: B

SUMMARY:
To compare in postmenopausal women with established osteoporosis the effect of treatment with teriparatide 20 micrograms/day subcutaneous with the effect of salmon calcitonin 100 IU/day subcutaneous on change in lumbar spine BMD.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, postmenopausal women aged 55-85 years (at least 3 years have elapsed after menopausal) are included at the time of entry into the trial. They have to be free of severe or chronically disabling conditions other than osteoporosis.
* The patient should have a documented (X-ray) prevalent osteoporotic vertebral fracture (defined as 3.4) or non vertebral fragility fracture (excluding major trauma).
* L-1 through L-4 vertebrae must be without artifacts, multiple vertebral fractures; therefore at least 3 vertebrae should be without fractures, osteophytes, or other abnormalities that would interfere with the analysis of the posterior-anterior lumbar spine BMD measurement. The reading of the BMD, T-score should be in the range of - 2.0 and - 4.0 at least for one of the 2 sites measured (spine or hip). The initial lumbar spine and femoral neck BMD assessment and the determination of the patient's eligibility for entry into the screening phase will be made by the central quality assurance for BMD. The central quality assurance center will determine the patient's eligibility for enrollment into the treatment phase. If the L-1 through L-4 vertebrae cannot be analyzed due to artifacts, vertebral fracture, osteophytes, or other abnormalities, that vertebra should be excluded from the analysis.
* Women without language barrier, cooperative expected to return for all follow-up procedures and who have given informed consent before entering the study and after being informed of the risks, medications, and procedures to be used in the study.
* Normal or clinically insignificant abnormal laboratory values including serum calcium, PTH(1-84) levels and alkaline phosphatase.

Exclusion Criteria:

* History of diseases which affect bone metabolism other than postmenopausal osteoporosis such as Paget's disease, renal osteodystrophy, osteomalacia, any secondary causes of osteoporosis, hypoparathyroidism, hyperparathyroidism, or hyperthyroidism.
* Patients who have an increased baseline risk of osteosarcoma: Paget's disease of the bone or unexplained elevations of alkaline phosphatase; Children and young adult with open epiphyses; Patients who have received radiation therapy involving the skeleton.
* History of other malignant neoplasms in the 5 years prior to screening, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated. Patients with carcinoma in situ of the uterine cervix treated definitively more than 1 year prior to entry into the study may enter the study.
* History of nephrolithiasis or urolithiasis in the 2 years prior to Visit 2. Patients with any history of nephro- or urolithiasis must have an appropriate radiology study within 6 months prior to Visit 2. This radiology study, such as an intravenous pyelogram or a supine radiograph of the kidney-ureter-bladder, must document the absence of active disease.
* History of sprue, inflammatory bowel disease, or malabsorption syndrome in the 1 year prior to Visit 2.

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-08; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
To compare in postmenopausal women with established osteoporosis the effect of treatment with teriparatide 20 micrograms/day subcutaneous with the effect of salmon calcitonin 100 IU/day subcutaneous on change in lumbar spine BMD.

SECONDARY OUTCOMES:
To compare in postmenopausal women with established osteoporosis the effect of treatment with teriparatide 20 micrograms/day with the effect of calcitonin 100 IU/day on change in femoral neck and total hip BMD
Compare effect of teriparatide 20 micrograms/day with the effect of calcitonin 100 IU/day on change in biochemical bone markers (bone specific alkaline phosphatase and Osteocalcin) at 3 and 6 months after treatment with teriparatide versus calcitonin.
Safety as determined by physical examinations, vital signs, clinical labs and reports of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMY - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com